CLINICAL TRIAL: NCT04962646
Title: CARbon Dioxide Flooding to Reduce Postoperative Neurological Injury Following Surgery for Acute Type A Aortic Dissection - A Prospective, Randomized, Blinded, Controlled Clinical Trial
Brief Title: CARbon Dioxide Flooding to Reduce Postoperative Neurological Injury Following Surgery for Acute Type A Aortic Dissection
Acronym: CARTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-02039
Record Dates: First submitted 2021-06-09; First posted 2021-07-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: D000784; D020521
Keywords: Aorta, Dissection, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, patient- and reviewer blinded interventional study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Once the thoracic cavity os opened during surgery, carbon dioxide flooding using a diffusor will be instigated with a flow of 5L/min. The flooding will be terminated once the aorta and the heart have no open contact with surrounding air.
  Interventions: Procedure: Carbon dioxide flooding
- Control (No Intervention): No intervention. No sham will be used as the staff performing the surgery would have been able to detect the lack of carbon dioxide in the surgical wound.

INTERVENTIONS:
Procedure: Carbon dioxide flooding — Once the thoracic cavity is opened a flow of carbon dioxide of 5L/min will be initiated into the surgical wound and proceed until there is no connection between the cardiac or aortic cavity and surrounding air.
  Arms: Intervention

SUMMARY:
Aortic dissection is a life-threatening condition and a consequence of a tear of the innermost of the three aortic layers- the intima. When a tear occurs, blood surges through the tear and causes the flow of blood between the aortic layers, causing a "false lumen". This causes a weakening of the aortic wall and hinders the blood from reaching its target organs and life saving emergent surgery is performed as routine.

Approximately 20% of patients undergoing acute type a aortic dissection (ATAAD) surgery suffer from postoperative neurological injuries and It has been demonstrated that neurological injuries account for 10-15% of in-hospital deaths.

In association with other cardiac procedures where the left side of the heart is opened and air may be trapped within the arterial circulation, carbon dioxide flooding is used to displace open air from the surgical wound. In comparison to air, carbon dioxide is significantly more soluble in blood and may therefore decrease the risk of air embolism. In cardiac surgery, carbon dioxide flooding has been demonstrated to reduce levels of biomarkers of cerebral injury, but carbon dioxide is not routinely employed in ATAAD surgery and has not been studied in association with these procedures.

The hypothesis is that carbon dioxide flooding reduces cerebral air embolism and the aim of this project is to evaluate whether carbon dioxide flooding may reduce neurological injuries following ATAAD surgery.

This is a prospective, randomized, controlled, patient- and reviewer blinded interventional study. Patients will be randomized to undergo surgery with carbon-dioxide flooding at 5L/min to the open chest cavity or conventional surgery without carbon dioxide flooding. Remaining aspects of the procedure will be identical.

The patient, external statistician and the reviewer analyzing the primary endpoints will be blinded for the randomization arms.

The study will assess the following endpoints:

Primary outcomes: Presence, number and volume of ischaemic lesions observed using magnetic resonance imaging (MRI) after ATAAD surgery.

Secondary outcomes: Clinical signs of neurological injury. Levels of biomarkers of neurological injury (S100B, neuron specific enolase (NSE) , neurofilament protein (NFL), Glial fibrillary acid protein (GFAP) , Ubiquitin carboxyl-terminal hydrolase L1 (UCH-L1) and Tau-protein (TAU)) before and after surgery. Quality of life, postoperative recovery and neurological function after ATAAD surgery. Primary outcomes in relation to retrograde cerebral perfusion.

Start of inclusion is anticipated to start Jan 1st, 2022. The writing of a manuscript describing the study methods and study objectives is expected to be started in 2021 and the final manuscript is expected to be written during 2025.

An interim analysis of the primary endpoints and the safety arm will be performed after 40 patients have been randomized. An external statistician together with the principle investigator will hereafter decide for the study to be continued or terminated due to harms, futility or superiority.

The safety arm will include intraoperative mortality, in-hospital mortality, re-operation for bleeding, stroke, myocardial infarction or other thromboembolic events.

Update August 2023:

Interim analyses were performed after 40 study participants had been included. Results from the interim analyses raised important questions which need to be assessed by a Data Safety and Monitoring Board (DSMB). Since there are no documented harmful effects of the intervention, a DSMB was not appointed before initiation of the trial. The study was suspended on Aug 18th 2023.

A DSMB will be appointed, analyze the interim analyses, collect necessary additional information and make a recommendation to the PI whether the study is may proceed or is to be terminated prematurely.

Update September 2023.

The DSMB has reviewed the interim analyses and additional study data. The DSMB concluded that there was no reason to terminate the study and have recommended for the study to proceed. Recruitment was re-initiated on September 5th 2023.

Update November 2024.

The study has recruited 68/80 participants. We anticipate that remaining participants will be recruited by June 2025.

ELIGIBILITY:
Inclusion Criteria:

* Verified acute type A aortic dissection.
* Patient accepted for surgical repair.

Exclusion Criteria:

* New-onset neurological symptoms defined as focal neurological symptoms or altered state of consciousness at time of inclusion.
* History of stroke with permanent neurological deficiency.
* Previous cardiac surgery.
* Surgery performed with cross clamping of the aorta without open distal anastomosis or open inspection of the distal aorta.
* Presence of implants or devices not compatible with Magnetic Resonance Imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of ischemic lesions on magnetic resonance imaging (MRI) | MRI will be performed before postoperative day 7. When not possible due to medical considerations, MRI may be performed up to 30 days after surgery.
  Number of ischemic lesions visualized using MRI
Size of ischemic lesions on magnetic resonance imaging (MRI) | MRI will be performed before postoperative day 7. When not possible due to medical considerations, MRI may be performed up to 30 days after surgery.
  Size of ischemic lesions visualized using MRI

SECONDARY OUTCOMES:
Clinical neurological injury | Up to postoperative day 7.
  Clinical neurological injury (Coma according to clinical neurological assessment and/or clinical focal neurological injuries assessed by neurologist or verified ischemic lesions on MRI).
Neurological function | Postoperative day 4 or at discharge from the ICU.
  Patients will be assessed using the National Institute of Health Stroke Scale (NIHSS). Minimum score 0 points, maximum score 42 points, with 42 points being the worst outcome.
Neurological function | Postoperative day 4 or at discharge from the ICU.
  Patients will be assessed using the modified Rankin Scale (mRS). Minimum score 0 points, maximum score 6 points, with 6 points being the worst outcome.
Level of consciousness | Postoperative day 4 or at discharge from the ICU.
  Patients will be assessed using the Glasgow Coma Scale Motor Score. Minimum score 1 points, maximum score 6 points, with 6 points being the best outcome.
Levels of S100B. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of S100B at predefined time points.
Levels of NSE. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of NSE at predefined time points.
Levels of NFL. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of NFL at predefined time points.
Levels of GFAP. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of GFAP at predefined time points.
Levels of UCH-L1. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of UCH-L1 at predefined time points.
Levels of TAU. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of TAU at predefined time points.
Neurological function after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the National Institute of Health Stroke Scale (NIHSS) three months after surgery. Minimum score 0 points, maximum score 42 points, with 42 points being the worst outcome.
Neurological function after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the modified Rankin Scale (mRS). Minimum score 0 points, maximum score 6 points, with 6 points being the best outcome.
Neurocognitive function after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the Symbol digit modalities test (SDMT). Minimum score 0 points, maximum score 110 points, with 110 points being the best outcome.
Cognitive function after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the Montereal cognitive assesment (MoCA) test. Minimum score 0 points, maximum score 30 points, with 30 points being the best outcome.
Neurological recovery after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the 2 simple questions for stroke). Minimum score 0 points, maximum score 2 points, with 2 points being the worst outcome.
Postoperative recovery after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the Postoperative recovery profile. Minimum score 19 points, maximum score 76 points, with 76 points being the best outcome.
Quality of life after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the Satisfaction with life scale. Minimum score 0 points, maximum score 35 points, with 35 points being the best outcome.
Quality of life after ATAAD surgery. | 3 months after surgery.
  Patients will be assessed using the EuroQol 5 dimensions 5 levels (EQ-5D-5L). Minimum score 5 points, maximum score 25 points, with 5 points being the best outcome.
Number of ischemic lesions on magnetic resonance imaging (MRI) in relation to the use of retrograde cerebral perfusion. | MRI will be performed before postoperative day 7. When not possible due to medical considerations, MRI may be performed up to 30 days after surgery.
  Number of ischemic lesions visualized using MRI analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Size of ischemic lesions on magnetic resonance imaging (MRI) in relation to the use of retrograde cerebral perfusion. | MRI will be performed before postoperative day 7. When not possible due to medical considerations, MRI may be performed up to 30 days after surgery.
  Size of ischemic lesions visualized using MRI analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of S100B analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of S100B at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of NSE analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of NSE at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of NFL analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of NFL at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of GFAP analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of GFAP at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of UCH-L1 analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of UCH-L1 at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.
Levels of TAU analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not. | Preoperatively, 24 hours from start of surgery, postoperative day 4 and 3 months after surgery.
  Concentration of TAU at predefined time points analysed in subgroups with patients that have received retrograde cerebral perfusion and those who have not.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zindovic, MD. PhD, Principal Investigator — Region Skåne, Skåne university hospital
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ede J, Teurneau-Hermansson K, Moseby-Knappe M, Ramgren B, Bjursten H, Ederoth P, Larsson M, Mattsson-Carlgren N, Sjogren J, Wierup P, Nozohoor S, Zindovic I. Carbon dioxide flooding to reduce postoperative neurological injury following surgery for acute type A aortic dissection: a prospective, randomised, blinded, controlled clinical trial, CARTA study protocol - objectives and design. BMJ Open. 2023 May 25;13(5):e063837. doi: 10.1136/bmjopen-2022-063837. PMID 37230515

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04962646/Prot_SAP_001.pdf